CLINICAL TRIAL: NCT00459537
Title: A Randomized, Open-label, Active-controlled, Multicenter, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of Topical 10% Terbinafine Hydrogen Chloride (HCl) Formulation Versus 5% Amorolfine Nail Lacquer for 48 Weeks of Treatment in Patients With Mild to Moderate Toenail Onychomycosis
Brief Title: Efficacy, Safety and Tolerability of Topical 10% Terbinafine Hydrogen Chloride Versus 5% Amorolfine Nail Lacquer in Patients With Mild to Moderate Toenail Onychomycosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSFO327N2303
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Onychomycosis
Keywords: Toenail fungus; Onychomycosis; Nail fungus; Toenail fungal infection; Tinea unguium; Dermatophytes; Foot dermatoses
MeSH Terms: conditions — Onychomycosis; Foot Dermatoses | interventions — Terbinafine

ARMS (2):
- Terbinafine (Experimental): 10% terbinafine hydrogen chloride (72.6 mg/ml nail lacquer). Patients applied one layer of the study medication once daily for 48 weeks, preferably at bedtime, to all affected toenails and allowed to dry.
  Interventions: Drug: terbinafine hydrogen chloride
- Amorolfine (Active Comparator): 5% amorolfine nail lacquer. Patients applied study medication twice weekly for 48 weeks to all affected toenails.
  Interventions: Drug: amorolfine nail lacquer

INTERVENTIONS:
Drug: terbinafine hydrogen chloride — 10 % terbinafine hydrogen chloride (HCL)
  Other Names: Lamisil
  Arms: Terbinafine
Drug: amorolfine nail lacquer — 5 % amorolfine nail lacquer
  Arms: Amorolfine

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of topical 10% terbinafine hydrogen chloride applied daily versus 5% amorolfine nail lacquer applied twice a week in patients with mild to moderate toenail onychomycosis, for a total treatment duration of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 12 - 75 years of age
* Fungal toenail infection of one or both of the large (great) toenails
* The nail infection must be due to a dermatophyte, (mixed infections [dermatophyte and non-dermatophyte] are not allowed)
* The target toenail area must have at least 25% to no more than 75% disease involvement without spikes.

Exclusion Criteria:

* Target foot must not have severe plantar (moccasin) tinea pedis that would require systemic therapy. Mild to moderate tinea pedis (athlete's foot) infection should be treated with terbinafine prior to baseline or at any time during the trial. Other topical treatments for athlete's foot may be recommended at the discretion of the investigator.
* Subjects must not have abnormalities of the nail that could prevent a normal appearing nail if clearing of infection is achieved
* No administration of systemic antifungal medications within 6 months prior to screening visit
* No application of prescription topical antifungal medications for toenail fungus within 3 months or other commercially available topical medications for toenail fungus applied directly to the toenails within 1 month prior to screening visit
* Patients with the target toenail involving the matrix (lunula) or having less than 2mm clear (unaffected) nail plate length beyond the proximal fold.
* Presence of dermatophytoma (defined as thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the target nail.
* No professional pedicures or application of any nail polish product or nail cosmetic to the toenails after the screening visit
* Known pregnancy or lactation at time of enrollment

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (10):
- Novartis Investigative Site, Various Cities, Finland
- Novartis Investigative Site, Various Cities, France
- Novartis Investigative Site, Various Cities, Germany
- Novartis Investigative Site, Various Cities, Hungary
- Novartis Investigative Site, Various Cities, Iceland
- Novartis Investigative Site, Various Cities, Norway
- Novartis Investigative Site, Various Cities, Poland
- Novartis Investigative Site, Various Cities, Russia
- Novartis Investigative Site, Various Cities, Spain
- Novartis Investigative Site, Various Cities, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Terbinafine | Amorolfine
Started | 507 | 522
Safety Population | 493 (Participants who had at least one dose of study drug and one post-baseline safety assessment.) | 512
Completed | 441 | 446
Not Completed | 66 | 76
Not completed — Adverse Event | 1 | 6
Not completed — Lack of Efficacy | 10 | 11
Not completed — Withdrawal by Subject | 20 | 26
Not completed — Lost to Follow-up | 27 | 30
Not completed — Administrative problems | 3 | 0
Not completed — Protocol Violation | 4 | 3
Not completed — Missing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Terbinafine | Amorolfine | Total
Number analyzed (Participants) | 507 | 522 | 1029
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 425 | 410 | 835
  >=65 years | 82 | 111 | 193
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 150 | 308
  Male | 349 | 372 | 721

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Cure at the End of Study After Treating Participants for 48 Weeks
Description: Complete cure is defined as negative potassium hydroxide (KOH) microscopy and negative culture for dermatophytes and no residual involvement of the target toenail.
Time Frame: Week 52
Population: The Intent-to-treat population (ITT) population consisted of all patients who were randomized and dispensed study drug. Last Observation Carried Forward (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Terbinafine | Amorolfine
Number analyzed (Participants) | 507 | 522
Percentage of participants | 1.18 | 0.96

2. Secondary Outcome: Percentage of Participants With Clinical Effectiveness at the End of Study After Treating Patients for 48 Weeks.
Description: Clinical effectiveness is defined as negative KOH microscopy and negative culture for dermatophytes and <= 10% residual involvement of the target toenail.
Time Frame: Week 52
Population: Intent-to-treat population, Last Observation Carried Forward (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Terbinafine | Amorolfine
Number analyzed (Participants) | 507 | 522
Percentage of participants | 4.54 | 3.83

3. Secondary Outcome: Percentage of Participants With Mycological Cure at End of Study After Treating Patients for 48 Weeks
Description: Mycological cure is defined as negative KOH microscopy and negative culture for dermatophytes
Time Frame: Week 52
Population: Intent-to-treat population, Last Observation Carried Forward (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Terbinafine | Amorolfine
Number analyzed (Participants) | 507 | 522
Percentage of participants | 16.17 | 15.71

4. Secondary Outcome: Safety and Tolerability Assessed by the Number of Participants With Adverse Events
Description: Safety and tolerability data as assessed by the number of participants with Adverse Events (AE), Serious Adverse Events, Drug discontinuation due to an AE or SAE and death. Additional details can be found in the Adverse Event Section.
Time Frame: Week 52
Population: The Safety population consisted of all patients that received at least one dose of study drug and had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Terbinafine | Amorolfine
Number analyzed (Participants) | 493 | 512
Participants
  At least 1 AE | 285 | 291
  AE suspected related to study drug | 11 | 7
  At least 1 SAE | 9 | 18
  SAE suspected related to study drug | 0 | 0
  Death | 0 | 0
  Drug discontinuation due to an AE | 1 | 5

5. Primary Outcome: Percentage of Participants With Complete Cure at the End of Study After Treating Participants for 48 Weeks.
Description: as for outcome 1
Time Frame: Week 52
Population: The Per-protocol population (PP) consisted of ITT patients who completed the study without protocol deviations that led to exclusion according to criteria defined before database lock The per-protocol population was used to provide confirmation of efficacy findings from the ITT population. Last Observation Carried Forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | Terbinafine | Amorolfine
Number analyzed (Participants) | 260 | 266
Percentage of participants | 1.15 | 0.38

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Safety population consisting of all patients who received at least one dose of study drug and had at least one post-baseline safety assessment.
Arm/Group | Terbinafine | Amorolfine
Serious Adverse Events (participants affected / at risk) | 9/493 | 18/512
Other Adverse Events (participants affected / at risk) | 186/493 | 168/512
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Terbinafine (N=493) | Amorolfine (N=512)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 1
Thyroid cyst (Endocrine disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Breast dysplasia (Reproductive system and breast disorders) | 0 | 1
Cyst removal (Surgical and medical procedures) | 1 | 0
Dupuytren's contracture operation (Surgical and medical procedures) | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Terbinafine (N=493) | Amorolfine (N=512)
Influenza (Infections and infestations) | 25 | 15
Nasopharyngitis (Infections and infestations) | 69 | 65
Tinea pedis (Infections and infestations) | 29 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 29
Headache (Nervous system disorders) | 98 | 70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.